CLINICAL TRIAL: NCT05608941
Title: Effects of High-Intensity Respiratory Muscle Training on Respiratory Muscle Strength, Functional Outcomes and Quality of Life in Individuals with Parkinson's Disease: a Randomized Clinical Trial
Brief Title: High-Intensity Respiratory Muscle Training in Individuals with Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Pró-reitoria de Pesquisa da Universidade Federal de Minas Gerais (Unknown)
Responsible Party: Principal Investigator, Christina Danielli Coelho de Morais Faria, Associate professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE: 53970421.0.0000.5149
Record Dates: First submitted 2022-10-27; First posted 2022-11-08 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease
Keywords: Breathing exercises; Clinical trial; Exercise; Muscle strength; Parkinson's disease; Rehabilitation
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Data collection and analysis will be carried-out by a researcher, blinded to the group allocation. In order to maintain the participants blinded to the training load, the device will be covered with opaque material.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): The training program will be carried-out with the Orygen Dual Valve. Individuals will perform a home-based intervention, split into two daily 20-min sessions (morning and afternoon), totaling 40 min per day, seven times a week, during eight weeks. Each daily session will be composed into four blocks of three minutes, with a two-minute rest between blocks. The initial training load for each participant will be set at 60% of his/her maximal baseline MIP and MEP for both inspiratory and expiratory strength training, respectively. Borg score of dyspnea and effort was also considered for adjusting training intensity, and scores from 4 to 6 were targeted. Once a week, a trained researcher will visit their homes, the MIP and MEP will be evaluated and the training load will be progressed to ensure that 60% of the new pressure values are maintained.
  Interventions: Other: Respiratory muscle training
- Control Group (Sham Comparator): The control group will also perform the exercises using the Orygen Dual Valve device. A sham intervention will be implemented: the initial resistance of the device will be 0cmH2O, and will be maintained throughout the intervention period - there will be no load progression. All procedures adopted with experimental group, including the weekly home visit, will also be performed with individuals in the control group. However, there will be no real change in the training load. All devices will be wrapped with an opaque material so that the load or possible respiratory training load is not visualized.
  Interventions: Other: Control

INTERVENTIONS:
Other: Respiratory muscle training — The training program will be carried-out with the Orygen Dual Valve. Individuals will perform a home-based intervention, split into two daily 20-min sessions (morning and afternoon), totaling 40 min per day, seven times a week, during eight weeks. Each daily session will be composed into four blocks of three minutes, with a two-minute rest between blocks. The initial training load for each participant will be set at 60% of his/her maximal baseline MIP and MEP for both inspiratory and expiratory strength training, respectively. Borg score of dyspnea and effort was also considered for adjusting training intensity, and scores from 4 to 6 were targeted. Once a week, a trained researcher will visit their homes, the MIP and MEP will be evaluated and the training load will be progressed to ensure that 60% of the new pressure values are maintained.
  Arms: Experimental Group
Other: Control — The control/sham group will underwent exactly the same protocol and weekly monitoring at home, but the participants will receive the devices without resistance of the spring.
  Arms: Control Group

SUMMARY:
Background: Individuals with PD commonly have a significant reduction in respiratory muscle strength and inspiratory muscle endurance, and it can intensify with the disease progression. Respiratory muscle training has shown to increase respiratory muscle strength in individuals with Parkinson's Disease (PD). However, the effect size on other functional outcomes has not been determined and/or investigated. In addition, no studies have investigated the effects of high-intensity respiratory muscle training (inspiratory and expiratory) in this population.

Objectives: The primary aim of this study will be to investigate the effects of high-intensity respiratory muscle training on inspiratory and expiratory muscle strength in individuals with PD. The secondary aim of this study will be to investigate the efficacy of high-intensity respiratory muscle training in improving inspiratory muscle endurance, peak cough flow, dyspnea, fatigue, exercise capacity, and quality of life in this population.

Design: A randomized controlled trial with blinded assessment will assign eligible participants to either: high-intensity respiratory muscle training (experimental group) or sham training (control group). Individuals will perform a home-based intervention, not directly supervised, consisted of two daily 20-min sessions (morning and afternoon), seven times a week, during eight weeks.

Study Outcomes: Primary outcomes are inspiratory and expiratory muscle strength (MIP and MEP). Secondary outcomes are respiratory muscle endurance, peak cough flow, dyspnea, fatigue, exercise capacity, and quality of life.The outcomes will be measured at baseline, post-intervention (after the 8-week intervention), and one month after the cessation of the intervention (12-week follow-up).

Conclusion: The results of this trial will provide valuable new information on the efficacy of high-intensity respiratory muscle training in improving muscle strength and other functional outcomes in individuals with PD.

DETAILED DESCRIPTION:
Sample size calculation: The sample size calculation was performed considering the primary outcome measures (inspiratory and expiratory muscle strength). The effect size for inspiratory muscle training was derived from a RCT with a similar population and intervention. Considering a significance level (α) of 5% and a power of 0.80, thirteen participants per group are required (a total of 26 participants). The effect size for expiratory muscle training was also derived from a RCT with a similar population and intervention. Considering a significance level (α) of 5% and a power of 0.80, fourteen participants per group are required (a total of 28 participants). Therefore, a sample size of 28 individuals (14 in each group) was defined (largest sample size calculated). Assuming an expected dropout rate of 20%, a total sample size of 34 individuals was set (17 in each group).

Statistical analyzes: All statistical analyzes will be performed by an independent examiner, blinded to the group allocation. Each participant will assigned a unique code. All analyzes will be performed using SPSS (SPSS Inc., Chicago, IL, USA). The normality of data distribution will be for all continuous numeric variables. Descriptive statistics will be calculated for all outcomes.The effects of the interventions will be analyzed from the collected data using intention-to-treat. Data from the last available assessment will be used for missed sessions. Two-way ANOVA with repeated measures (2*3) will be used to evaluate the differences between groups, considering the time factor (considering baseline, post-intervention, and 4-week follow-up), for the variables: inspiratory and expiratory muscle strength, respiratory muscle endurance, peak cough flow and exercise capacity. The level of significance will be set at 5% and adjusted for multiple comparisons. Data distribution and equality of variance will also be analyzed, to ensure the parametric analysis has been applied correctly. The effect sizes will be calculated to determine the magnitude of the differences between the groups. The differences between the two mean values will be expressed in units of their SD, expressed as Cohen's d, or mean results for the experimental group minus the mean results for the control group, divided by the SD of the control group. Effect sizes between 0.2 and 0.5 will be considered small; between 0.5 and 0.8, medium; and above 0.8, large.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease diagnosed by a neurologist
* Ability to walk independently, with or without assistive devices
* Taking anti parkinsonian medication, and who have been medically stable for at least six months
* Classified between stages 1-3 of the modified Hoehn & Yahr Scale (Schenkman et al., 2001)
* Maximum inspiratory pressure less or equal to -80 cmH2O or maximum expiratory pressure less or equal to 90 cmH2O

Exclusion Criteria:

* Possible cognitive impairment as determined by cutoff scores (in points) of the Mini-Mental Status Examination
* Use deep brain stimulation (DBS)
* Smokers or who stopped smoking less than six months ago; have been affected by respiratory or cardiac infections in the last month
* Had any other neurological, musculoskeletal, cardiovascular or respiratory disorders that could affect their ability to perform the tests

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Maximal inspiratory pressure (MIP) | At baseline, post-intervention (after the 8-week intervention), and one month after the cessation of the intervention (12-week follow-up).
  Maximum inspiratory pressure will be measured using a digital manovacuometer (LEB-LabCare/UFMG, Brazil) , following previously described protocols.
Change from baseline in Maximal expiratory pressure (MEP) | At baseline, post-intervention (after the 8-week intervention), and one month after the cessation of the intervention (12-week follow-up).
  Maximum expiratory pressure will be measured using a digital manovacuometer (LEB-LabCare/UFMG, Brazil) , following previously described protocols.

SECONDARY OUTCOMES:
Change from baseline in Inspiratory muscle endurance | At baseline, post-intervention (after the 8-week intervention), and one month after the cessation of the intervention (12-week follow-up).
  Inspiratory endurance will be assessed by the powerbreathe device. The measurement will be carried out following the recommended guideline for the flow-resistive loading tests.
Change from baseline in Peak cough flow | At baseline, post-intervention (after the 8-week intervention), and one month after the cessation of the intervention (12-week follow-up).
  Peak cough flow measurement will be performed with the with peak expiratory flow meter (Mini-Wright Peak Expiratory Flow Meter), following previously described protocols.
Change from baseline in perception of Dyspnea | At baseline, post-intervention (after the 8-week intervention), and one month after the cessation of the intervention (12-week follow-up).
  Dyspnea will be measured using the instrument of the Medical Research Council (MRC). This is a 5-point scale, in which 0 indicates 'breathless only with strenuous exercise' and 4 indicates 'too breathless to leave the house'.
Change from baseline in Fatigue | At baseline, post-intervention (after the 8-week intervention), and one month after the cessation of the intervention (12-week follow-up).
  Fatigue will be measured using the Fatigue Severity Scale. The scale consists of 9 items, for each item the scores range from 1 (strongly disagree) to 7 (strongly agree). A higher score indicates a higher level of fatigue.
Change from baseline in Exercise capacity | At baseline, post-intervention (after the 8-week intervention), and one month after the cessation of the intervention (12-week follow-up).
  Exercise capacity will be measured using the Six-minute Walk Test (6MWT), following previously described protocols.
Change from baseline in Quality of life | At baseline, post-intervention (after the 8-week intervention), and one month after the cessation of the intervention (12-week follow-up).
  Quality of life will be measured using the Parkinson's Disease Questionnaire-39. This instrument is composed of 39 items divided into eight dimensions. The score for each domain ranges from 0 (zero) to 100 (one hundred), where zero means better and one hundred means worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Christina CM Faria, Doctor, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brito SAF, Scianni AA, Silveira BMF, Oliveira ERM, Mateus ME, Faria CDCM. Effects of high-intensity respiratory muscle training on respiratory muscle strength in individuals with Parkinson's disease: Protocol of a randomized clinical trial. PLoS One. 2023 Sep 8;18(9):e0291051. doi: 10.1371/journal.pone.0291051. eCollection 2023. PMID 37682839